CLINICAL TRIAL: NCT03619811
Title: Precision Approach to PPI Therapy in Gastroesophageal Reflux Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Rena Yadlapati, Principal Investigator, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18-0205
Record Dates: First submitted 2018-07-19; First posted 2018-08-08 (Actual); Results first posted 2021-09-20 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-08

CONDITIONS: Gastroesophageal Reflux; Laryngopharyngeal Reflux
Keywords: esophageal disorders
MeSH Terms: conditions — Gastroesophageal Reflux; Laryngopharyngeal Reflux; Esophageal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Symptomatic (Experimental): This study examines the efficacy of the upper esophageal sphincter assist device as an adjunct to Proton-pump inhibitors (PPI) therapy in symptomatic subjects. (Reflux Band® Upper Esophageal Sphincter (UES) Assist Device)
  Interventions: Diagnostic Test: Reflux Band® Upper Esophageal Sphincter (UES) Assist Device

INTERVENTIONS:
Diagnostic Test: Reflux Band® Upper Esophageal Sphincter (UES) Assist Device — UES augmentation via the UES assist device is effective in true Reflux associated laryngeal symptoms. In our first pilot trial with the UES assist device, patients had significant symptom reduction following 2 weeks of UES assist device use. Based on our preliminary work, we theorize that the UES assist device is effective in Reflux associated laryngeal symptoms.

SUMMARY:
This study plans to learn more about reflux associated laryngeal symptoms, and more efficient ways to diagnose and treat this condition.

DETAILED DESCRIPTION:
Reflux associated laryngeal symptoms, coined "laryngopharyngeal reflux", occurs when gastro-esophago-pharyngeal reflux contributes to chronic laryngeal symptoms such as throat clearing, sore throat and dysphonia. Over the past 25 years, Reflux associated laryngeal symptoms has been increasingly, and often incorrectly, diagnosed and has emerged as a point of controversy and confusion.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-89 years male and female,
* >8 weeks of symptoms of sore throat, throat clearing, and/or voice hoarseness,
* naïve to PPI or able to stop for 8 weeks

Exclusion Criteria:

* Laryngeal mass lesion on laryngoscopy;
* Pregnant;
* Unable to consent in English;
* Imprisoned;
* PPI intolerance;
* Contraindication to UESAD use per manufacturer guidelines which include:

  * Patients with implants or implant parts that reside in the area where UESAD is applied.
  * Patients with an implanted pacemaker, implanted cardioverter defibrillator (ICD), vagus nerve stimulator, or other such similar devices implanted in the neck.
  * Patients diagnosed with glaucoma.
  * Patients who had a malignancy of the neck, including neck surgery.
  * Patients that may have an altered mental status including due to the use of sedative drugs or narcotics.
  * Patients with carotid artery disease, thyroid disease, a history of cerebrovascular disease, or any disorder of connective tissues (e.g., Marfan's Syndrome or Ehlers-Danlos Syndrome).
  * Patients who use nocturnal NIV machines such as CPAP or BiPAP.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2018-07-13 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rena Yadlapati, M.D., Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yadlapati R, Pandolfino JE, Greytak M, Cahoon J, Clarke M, Clary M, Fink D, Menard-Katcher P, Vahabzadeh-Hagh AM, Weissbrod P, Gupta S, Kaizer A, Wani S. Upper Esophageal Sphincter Compression Device as an Adjunct to Proton Pump Inhibition for Laryngopharyngeal Reflux. Dig Dis Sci. 2022 Jul;67(7):3045-3054. doi: 10.1007/s10620-021-07172-2. Epub 2021 Jul 18. PMID 34275061

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Symptomatic
Started | 43
Completed | 31
Not Completed | 12

BASELINE CHARACTERISTICS:
Arm/Group | Symptomatic
Number analyzed (Participants) | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 33
  >=65 years | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.48 (15.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White / Caucasian | 26
  Black | 1
  Asian | 2
  Hispanic | 10
  Other | 4
Region of Enrollment [Number; unit: participants]
  United States | 43
Reflux Symptom Index Baseline [Mean (Standard Deviation); unit: units on a scale] | 24.1 (10.9)

OUTCOME MEASURES:

1. Primary Outcome: Patient-reported Symptom Response to Treatment Measured by the Reflux Symptom Index (RSI) Score
Description: Response will be assessed binary as positive or negative where a positive response is defined by a post-treatment reflux symptom index (RSI) score ≤ 13 and a 33% change from comparator RSI. The minimum value is 0 and the maximum value is 45. The lower the score means less reported symptoms and the higher the score means more reported symptoms.
Time Frame: Week 8 (Completion)
Population: This analysis includes the participants that completed phase 1 & 2 of the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Symptomatic
Number analyzed (Participants) | 31
score on a scale | 15.5 (10.3)

2. Primary Outcome: Patient-reported Symptom Response to Treatment Measured by the Reflux Symptom Index (RSI) Score
Description: as for outcome 1
Time Frame: Week 4
Population: This population completed phase 1.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Symptomatic
Number analyzed (Participants) | 36
score on a scale | 21.9 (9.7)

ADVERSE EVENTS:
Time Frame: 26 months
Description: Standard definitions of adverse event and/or serious adverse event were used to collect adverse event information.
Arm/Group | Symptomatic
All-Cause Mortality (participants affected / at risk) | 0/43
Serious Adverse Events (participants affected / at risk) | 0/43
Other Adverse Events (participants affected / at risk) | 1/43
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Symptomatic (N=43)
Discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) — Collar bone discomfort reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-30): https://cdn.clinicaltrials.gov/large-docs/11/NCT03619811/Prot_SAP_000.pdf